CLINICAL TRIAL: NCT03387059
Title: A Multicentre, Prospective Randomised Controlled, Interventional Clinical Investigation to Assess the Clinical Safety and Performance of Forielle, a Medical Device for Endometrial Washing in Restoring Favorable Endometrial Condition to Implantation After COS During Assisted Reproductive Practice (ENDOMEDE)
Brief Title: Clinical Performance and Safety Investigation of ENDOmetrial Washing MEdical DEvice Forielle
Acronym: ENDOMEDE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated early, due to the poor feasibility and sustainability, leading to slow recruitment rate.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.P.A., Italy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS700623-0009
Record Dates: First submitted 2017-12-22; First posted 2017-12-29 (Actual); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-08

CONDITIONS: Infertility
Keywords: Infertility; Forielle; Assisted Reproductive Technique (ART); Controlled Ovarian Stimulation (COS)
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forielle Endometrial Washing (Experimental)
  Interventions: Device: Forielle
- No Endometrial Washing (No Intervention)

INTERVENTIONS:
Device: Forielle — Participants randomized to receive Forielle endometrial washing (an intrauterine solution) following oocyte retrieval on Study Day 0 (Randomisation).
  Arms: Forielle Endometrial Washing

SUMMARY:
This is a multicenter, prospective randomized controlled, interventional investigation to assess the safety and clinical performance of Forielle, a medical device for endometrial washing, in restoring favorable endometrial condition to implantation after Controlled Ovarian Stimulation (COS) during Assisted Reproductive Technique (ART).

ELIGIBILITY:
Inclusion Criteria:

* All infertile women treated with intracytoplasmic sperm injection (ICSI)/Fertilization in Vitro and Embryo Transfer (FIVET)
* Less than or equal to (<=) 1 previous failed embryo transfer
* Eumenorrheic normo-gonadotropic women
* Basal follicle-stimulating hormone (FSH) <=12 International unit per liter (IU/L)
* Anti-mullerian hormone (AMH) greater than (>) 1.1 nanogram per milliliter (ng/mL)
* Ovarian Reserve: number of antral follicles 2 millimeter (mm) between 6 <= antral follicle count (AFC) <= 16
* Follicles > 16 mm at the triggering day between 5-14
* Body Mass Index (BMI) between 18 <= BMI <= 27 kilogram per meter square (kg/m^2)
* Indication for Fresh Embryo transfer
* Normal uterine cavity on ultrasound exam (e.g., no presence of hydrosalpinx)
* Undergoing Assisted Reproductive Technique (ART) and oocyte maturation by human chorionic gonadotropin (HCG) triggering
* Progesterone (P4) serum level at the HCG triggering day <= 1.5 ng/mL (Day O/Randomization)
* Estradiol (E2) <= 3000 picogram/milliliter (pg/mL) at the human chorionic gonadotropin (HCG) triggering day (Day 0/Randomization)
* Subjects must have read and signed the Informed Consent Form prior to study-specific-procedures not part of standard of care
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Clinically significant systemic disease (such as diabetes, metabolic syndrome, immunological diseases, diagnosed thrombophilia, porphyria, or any other medical condition requiring the use of low-molecular weight heparin therapy)
* Polycystic ovary syndrome (PCOS) according to Rotterdam Consensus Criteria (European Society of Human Reproduction and Embryology [ESHRE]/American Society for Reproductive Medicine [ASRM], 2003)
* Poor ovarian response (POR) according to the European Society of Human Reproduction and Embryology (ESHRE) Criteria
* RIF (repeated implantation failure), defined as greater than or equals to (>=) 2 previous failed embryo transfers
* Endometriosis III-IV stage or adenomyosis
* Clinically significant findings on exam or ultrasound, such as salpingitis, hydrosalpynx or evidence of ovarian cysts
* Known hypersensitivity to any of the components of the solution
* Known hypersensitivity to vaginal progesterone or its excipients
* Other protocol defined exclusion criteria could apply

Max Age: 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (7):
- Italy (7):
  - Unità Operativa di Fisiopatologia della Riproduzione - Ospedale Cervesi di Cattolica, Cattolica
  - Centro di Procreazione Assistita Demetra, Florence
  - Centro di Procreazione Medicalmente Assistita - Ospedale di Versilia, Lucca
  - Humanitas Fertility Center, Milan
  - Centro Scienze della Natalità - IRCCS Ospedale San Raffaele, Milan
  - Unità Operativa di Ginecologia - Istituti Clinici Zucchi, Monza
  - Centro di Procreazione Medicalmente Assistita (PMA) - Casa di Cura PROMEA, Torino

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Nine participants were enrolled and the study was prematurely terminated due to the poor feasibility and sustainability, leading to slow recruitment rate.
Groups:
- Forielle Endometrial Washing: Participants randomized in this group were assessed using Forielle endometrial washing (an intrauterine solution) following oocyte retrieval on Study Day 0 (Randomization).
- No Endometrial Washing: Participants randomized in this group (Control) were assessed without using Forielle endometrial washing (an intrauterine solution) following oocyte retrieval on Study Day 0 (Randomization).
Period: Overall Study
Arm/Group | Forielle Endometrial Washing | No Endometrial Washing
Started | 5 | 4
Completed | 0 | 0
Not Completed | 5 | 4
Not completed — Study termination | 5 | 4

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all randomized participants into the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Forielle Endometrial Washing | No Endometrial Washing | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Implantation Rate
Description: Implantation rate was defined as the number of intrauterine gestational sacs divided by the number of embryos transferred.
Time Frame: Post Embryo Transfer (PET) Days 21 to 28
Population: Data was not collected since the study was terminated early due to the poor feasibility and sustainability, leading to slow recruitment rate.
Arm/Group | Forielle Endometrial Washing | No Endometrial Washing
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants With Positive and Negative Pregnancy
Description: Positive and Negative Pregnancy measured by Day 14 serum beta Human chorionic gonadotropin (Beta-HCG) pregnancy test.
Time Frame: At Post Embryo Transfer (PET) Day 14
Population: as for outcome 1
Arm/Group | Forielle Endometrial Washing | No Endometrial Washing
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Confirmed Ongoing Pregnancy
Description: Ongoing pregnancy was defined as having a positive fetal heart beat (FHB) as assessed by obstetric ultrasound (transvaginal or abdominal).
Time Frame: Post Embryo Transfer (PET) Days 70 to 84
Population: as for outcome 1
Arm/Group | Forielle Endometrial Washing | No Endometrial Washing
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Device Incidents
Description: A medical device incident is any malfunction or deterioration in the characteristics and/or clinical performance of a device, as well as any inadequacy in the labelling or the instructions for use (IFU) which, directly or indirectly, might lead to or might have led to the death of a participant, or user or of other persons or to a serious deterioration in their state of health.
Time Frame: Day 2 post-randomization (PR) up to Post Embryo Transfer (PET) Days 70 to 84
Population: as for outcome 1
Arm/Group | Forielle Endometrial Washing | No Endometrial Washing
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 152
Arm/Group | Forielle Endometrial Washing | No Endometrial Washing
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

LIMITATIONS AND CAVEATS:
The study was terminated early, due to the poor feasibility and sustainability, leading to slow recruitment rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT03387059/Prot_SAP_000.pdf